CLINICAL TRIAL: NCT05330455
Title: Four-part, Randomized, Double-blind (Parts 1, 2A, 3 and 4), Multi-center, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSK3965193 Monotherapy in Healthy Participants and in Participants Living With Chronic Hepatitis B Infection; and GSK3965193 in Combination With Bepirovirsen in Participants Living With Chronic Hepatitis B Infection
Brief Title: Study of GSK3965193 in Healthy Participants and Participants Living With Chronic Hepatitis B Infection
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 214760; 2021-005117-13 (EudraCT Number); 2023-509684-24 (Other: EU CTR)
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Hepatitis B
Keywords: Bepirovirsen; Chronic hepatitis B; First-time-in-human; GSK3965193
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic

STUDY DESIGN:
Intervention Model Description: Parts 1 and Part 2B are crossover and Part 2A, Part 3 and Part 4 are parallel group
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Part 1 Cohort 1: GSK3965193 and placebo (Experimental): Healthy participants will be randomized to receive single ascending doses of GSK3965193 and placebo in one of 4 treatment sequences in a 3:1 ratio in fasted conditions. In period 1, participants will receive GSK3965193 (Dose 1) + Placebo; in period 2: GSK3965193 (Dose 2) + Placebo; in period 3: GSK3965193 (Dose 3) + Placebo and in period 4: GSK3965193 (Dose 4) + Placebo. There will be a minimum of 7 days washout between dosing in each treatment period.
  Interventions: Drug: GSK3965193; Drug: Placebo to match GSK3965193
- Part 1 Cohort 2: GSK3965193 and placebo (Experimental): Healthy participants will be randomized to receive single ascending doses of GSK3965193 and placebo in one of 4 treatment sequences in a 3:1 ratio in fasted conditions. In period 1, participants will receive GSK3965193 (Dose 5) + Placebo; in period 2: GSK3965193 (Dose 6) + Placebo; in period 3: GSK3965193 (Dose 7) + Placebo and in period 4: GSK3965193 (Dose 8) + Placebo. There will be a minimum of 7 days washout between dosing in each period.
  Interventions: Drug: GSK3965193; Drug: Placebo to match GSK3965193
- Part 2A Cohort 3: GSK3965193 or placebo (Experimental): Healthy participants will be randomized 3:1 to receive repeat doses of either GSK3965193 (Dose X) or placebo under fasted conditions. Part 2A may start while Part 1 is still ongoing. The starting dose in Part 2 will be at least 3-fold below the highest dose completed in Part 1.
  Interventions: Drug: GSK3965193; Drug: Placebo to match GSK3965193
- Part 2A Cohort 4: GSK3965193 or placebo (Experimental): Healthy participants will be randomized 3:1 to receive repeat doses of either GSK3965193 (Dose X) or placebo under fasted conditions. Part 2A may start while Part 1 is still ongoing. The starting dose in Part 2 will be at least 3-fold below the highest dose completed in Part 1.
  Interventions: Drug: GSK3965193; Drug: Placebo to match GSK3965193
- Part 2A Cohort 5: GSK3965193 or placebo (Experimental): Healthy participants will be randomized 3:1 to receive repeat doses of either GSK3965193 (Dose X) or placebo under fasted conditions. Part 2A may start while Part 1 is still ongoing. The starting dose in Part 2 will be at least 3-fold below the highest dose completed in Part 1.
  Interventions: Drug: GSK3965193; Drug: Placebo to match GSK3965193
- Part 2B Cohort 6: GSK3965193 (Experimental): Healthy Participants will be randomized 1:1 to receive single doses of GSK3965193 (Dose A) under fasted and fed conditions in treatment period 1. In period 2, the participants who received GSK3965193 (Dose A) under fasted conditions in treatment period 1 will receive the same dose under fed conditions, and vice versa. In the third period, all participants will receive a single dose of GSK3965193 (Dose B) different strength under fasted conditions. The dose level for the third period will be selected based on the results of the first two periods. There will be a minimum of 7 days washout between dosing in each treatment period.
  Interventions: Drug: GSK3965193
- Part 3 Cohort 7: GSK3965193 or placebo (Experimental): PLWCHB on stable nucleos(t)ide analog (NA) therapy will be randomized 3:1 to receive repeat dose of either GSK3965193 (Dose E) or placebo. This part will commence after completion of both Part 1 and Part 2.
  Interventions: Drug: GSK3965193; Drug: Placebo to match GSK3965193
- Part 3 Sub-Cohort 7: Open label bepirovirsen (Experimental): PLWCHB participants on stable NA therapy who have completed GSK3965193/placebo monotherapy (Part 3, Cohort 7) will be given the option to receive subsequent treatment of optional open label bepirovirsen only for 24 weeks.
  Interventions: Drug: Bepirovirsen
- Part 4 Cohort 8: GSK3965193 and bepirovirsen or placebo and bepirovirsen (Experimental): PLWCHB participants on stable NA therapy who have not participated in Part 3 of the study will be randomized 3:1 to receive repeat dose either GSK3965193 or placebo. In addition, all participants in this cohort will also receive bepirovirsen. This part will commence after completion of Part 3, contingent on the clinical safety and efficacy data from Part 3.
  Interventions: Drug: GSK3965193; Drug: Placebo to match GSK3965193; Drug: Bepirovirsen

INTERVENTIONS:
Drug: GSK3965193 — GSK3965193 will be administered
  Arms: Part 1 Cohort 1: GSK3965193 and placebo; Part 1 Cohort 2: GSK3965193 and placebo; Part 2A Cohort 3: GSK3965193 or placebo; Part 2A Cohort 4: GSK3965193 or placebo; Part 2A Cohort 5: GSK3965193 or placebo; Part 2B Cohort 6: GSK3965193; Part 3 Cohort 7: GSK3965193 or placebo; Part 4 Cohort 8: GSK3965193 and bepirovirsen or placebo and bepirovirsen
Drug: Placebo to match GSK3965193 — Placebo to match GSK3965193 will be administered
  Arms: Part 1 Cohort 1: GSK3965193 and placebo; Part 1 Cohort 2: GSK3965193 and placebo; Part 2A Cohort 3: GSK3965193 or placebo; Part 2A Cohort 4: GSK3965193 or placebo; Part 2A Cohort 5: GSK3965193 or placebo; Part 3 Cohort 7: GSK3965193 or placebo; Part 4 Cohort 8: GSK3965193 and bepirovirsen or placebo and bepirovirsen
Drug: Bepirovirsen — Bepirovirsen will be administered
  Arms: Part 3 Sub-Cohort 7: Open label bepirovirsen; Part 4 Cohort 8: GSK3965193 and bepirovirsen or placebo and bepirovirsen

SUMMARY:
This Phase 1/2a multiple part study is a first time-in-human (FTIH) study designed to evaluate the safety, tolerability, and pharmacokinetics (PK) of single (Part 1) and repeat doses (Part 2) of GSK3965193 in healthy participants. Part 3 will evaluate the ability of GSK3965193 to lower hepatitis B virus surface antigen (HBsAg) in participants living with chronic hepatitis B infection (PLWCHB) and will be given the option to subsequently receive treatment with open label bepirovirsen. Part 4 will evaluate the safety and tolerability of combination therapy with GSK3965193 and bepirovirsen and the potential to effect sustained virologic response in PLWCHB.

ELIGIBILITY:
Inclusion Criteria:

Parts 1 and 2: Participants between 18 and 55 years of age inclusive, at the time of signing the informed consent.

* Parts 3 and 4: Participants between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Body weight >=50 kilograms (kg) and body mass index within the range 18-32 kilograms per square meter (kg/m^2) (inclusive).
* Male or female participant: a. Parts 1 and 2: woman of nonchildbearing potential only. b. Parts 3 and 4: woman of nonchildbearing potential or woman of child-bearing potential who is not pregnant or breastfeeding and is using a contraceptive method that is highly effective.
* Capable of giving signed informed consent.
* Additional Inclusion Criteria for PLWCHB (Parts 3 and 4).
* Participants who have documented chronic hepatitis B virus (HBV) infection >=6 months prior to screening.
* Participants currently receiving stable NA therapy (e.g., tenofovir disoproxil, tenofovir alafenamide, entecavir).
* Plasma or serum HBsAg concentration >100 IU/mL.
* Plasma or serum HBV deoxyribonucleic acid (DNA) concentration <90 IU/mL.
* Hepatitis B virus e-antigen (HBeAg) positive or negative.
* Alanine aminotransferase (ALT) <=2 times the upper limit of normal (ULN)

Exclusion Criteria:

Exclusion Criteria for Healthy Participants:

* Positive Hepatitis A virus antibody (HAV Ab immunoglobulin M [IgM]), or positive for HBV, hepatitis C virus (HCV) or human immunodeficiency virus (HIV) at screening
* A current diagnosis of migraine headache
* ALT >1 times ULN.
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%])
* Corrected QT interval (QTc) >450 milliseconds (msec)
* Signs and symptoms suggestive of Coronavirus Disease 2019 (COVID-19)
* Participants with known COVID-19 positive contacts in the past 14 days.
* For participants in Part 2A: i. Personal history or family history of peripheral neuropathy. ii. A score ≥4 on the Toronto clinical scoring system for polyneuropathy
* Current or previous use of tobacco- or nicotine-containing products (for example (e.g.) cigarettes, nicotine patches or electronic devices) within 6 months before screening and/or have a smoking pack history of >5 pack years

Exclusion Criteria for PLWCHB:

* Clinically significant abnormalities affecting physical or mental health in medical history or on physical examination, aside from chronic HBV infection.
* Co-infection with or past history of HCV, HIV or Hepatitis D virus (HDV).
* History of or suspected liver cirrhosis and/or evidence of cirrhosis.
* Diagnosed or suspected hepatocellular carcinoma.
* History of malignancy within the past 5 years with the exception of specific cancers that are cured by surgical resection (e.g., skin cancer).
* History of vasculitis or presence of symptoms and signs of potential vasculitis [e.g., vasculitic rash, skin ulceration, repeated blood detected in urine without identified cause] or history/presence of other diseases Exclusion Criteria for Healthy Participants:
* Positive Hepatitis A virus antibody (HAV Ab immunoglobulin M [IgM]), or positive for HBV, hepatitis C virus (HCV) or human immunodeficiency virus (HIV) at screening.
* A current diagnosis of migraine headache
* ALT >1 times ULN.
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]).
* Corrected QT interval (QTc) >450 milliseconds (msec).
* Signs and symptoms suggestive of Coronavirus Disease 2019 (COVID-19).
* Participants with known COVID-19 positive contacts in the past 14 days.
* For participants in Part 2A: i. Personal history or family history of peripheral neuropathy. ii. A score ≥4 on the Toronto clinical scoring system for polyneuropathy.
* Current or previous use of tobacco- or nicotine-containing products (for example (e.g.) cigarettes, nicotine patches or electronic devices) within 6 months before screening and/or have a smoking pack history of >5 pack years

Exclusion Criteria for PLWCHB:

* Clinically significant abnormalities affecting physical or mental health in medical history or on physical examination, aside from chronic HBV infection.
* Co-infection with or past history of HCV, HIV or Hepatitis D virus (HDV).
* History of or suspected liver cirrhosis and/or evidence of cirrhosis.
* Diagnosed or suspected hepatocellular carcinoma.
* History of malignancy within the past 5 years with the exception of specific cancers that are cured by surgical resection (e.g., skin cancer).
* History of vasculitis or presence of symptoms and signs of potential vasculitis [e.g., vasculitic rash, skin ulceration, repeated blood detected in urine without identified cause] or history/presence of other diseases that may be associated with vasculitis condition (e.g., systemic lupus erythematosus, rheumatoid arthritis, relapsing polychondritis, mononeuritis multiplex).
* History of extrahepatic disorders possibly related to HBV immune conditions (e.g., nephrotic syndrome, any type of glomerulonephritis, polyarteritis nodosa, cryoglobulinaemia, uncontrolled hypertension).
* History of alcohol or drug abuse/dependence: a. Current alcohol use as judged by investigator to potentially interfere with participant compliance. b. History of or current drug abuse/dependence as judged by the investigator to potentially interfere with participant compliance.
* History or other evidence of bleeding from esophageal varices.
* Documented history or other evidence of metabolic liver disease within 1 year of randomization.
* Personal history or family history of peripheral neuropathy.
* A score >4 on the Toronto clinical scoring system for polyneuropathy.
* History of having received or currently receiving any systemic anti-neoplastic (including radiation) or immune-modulatory treatment (including systemic oral corticosteroids, interferon or pegylated interferon) within the 3 months prior to randomization or the expectation that such treatment will be needed at any time during the study.
* Abnormal and clinically significant 12-lead ECG finding.
* Currently taking, or taken within 3 months prior to randomization, any immunosuppressing drugs (e.g., prednisone), other than a short course of therapy (≤2 weeks) or topical/inhaled steroid use.
* Participants requiring anti-coagulation therapies.
* Prior treatment with any oligonucleotide or small interfering RNA (siRNA) within 12 months prior to the first dosing day.
* Positive test for COVID-19 infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Parts 1 and 2B: Number of participants with adverse events (AEs), serious adverse events (SAEs), and withdrawals due to AEs | Up to 14 days
Part 2A: Number of participants with AEs, SAEs, and withdrawals due to AEs | Up to 42 Days
Parts 1: Number of participants with clinically significant changes in laboratory parameters | Up to 2 days
Parts 2B: Number of participants with clinically significant changes in laboratory parameters | Up to 14 days
Parts 1 and 2B: Number of participants with clinically significant changes in vital signs and cardiac parameters (electrocardiogram [ECG]) | Up to 14 days
Part 2A: Number of participants with clinically. significant changes in laboratory parameters, vital signs, cardiac parameters (ECG) | Up to 21 days
Part 2A: Number of participants with clinically. significant nerve changes | Up to 42 days
Part 1 and 2B: Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-inf]) of GSK3965193 following single dose administration | Up to 4 days
Part 2A: AUC(0-tau) of GSK3965193 following repeat dose administration | Up to 17 days
Part 1 and 2B: maximum observed concentration (Cmax) of GSK3965193 following single dose administration | Up to 4 days
Part 2A: Cmax of GSK3965193 following repeat dose administration | Up to 17 days
Part 1 and 2B: Time to maximum observed plasma drug concentration (Tmax) of GSK3965193 following single dose administration | Up to 4 days
Part 2A: Tmax of GSK3965193 following repeat dose administration | Up to 17 days
Part 1 and 2B: Apparent terminal half-life (T1/2) of GSK3965193 following single dose administration | Up to 4 days
Part 2A: T1/2 of GSK3965193 following repeat. dose administration | Up to 17 days
Part 3: Number of participants with AEs, SAEs, and withdrawals due to AEs | Up to 42 days
Part 4: Number of participants with AEs, SAEs, and withdrawals due to AEs | Up to 48 weeks
Part 3: Number of participants with clinically. significant changes in laboratory parameters and vital signs | Up to 42 days
Part 3: Number of participants with clinically. significant changes in cardiac parameters (ECG) | Up to 42 days
Part 4: Number of participants with clinically. significant changes in laboratory parameters and vital signs | Up to 48 weeks
Part 4: Number of participants with clinically. significant changes in cardiac parameters (ECG) | Up to 48 weeks
Part 3: Number of participants with clinically. significant nerve changes | Up to 42 days
Part 4: Number of participants with clinically. significant nerve changes | Up to 48 weeks
Part 3: Maximum reduction of serum HBsAg levels from Baseline | Baseline and up to 6 weeks
Part 4: Number of participants achieving. complete response | Up to 48 weeks

SECONDARY OUTCOMES:
Part 2B: AUC (0-inf) of GSK3965193 following. single dose administration | Up to 4 days
Part 2B: Cmax of GSK3965193 following single dose administration | Up to 4 days
Part 3: AUC(0-tau) of GSK3965193 following. repeat dose administration | Up to 42 days
Part 3: Cmax of GSK3965193 following repeat dose administration | Up to 42 days
Part 3: Tmax of GSK3965193 following repeat. dose administration | Up to 42 days
Part 3: T1/2 of GSK3965193 following repeat. dose administration | Up to 42 days
Part 3: Change from baseline in serum HBsAg levels from baseline (greater than or equal to [≥] 0.5 times log international units per milliliters [IU/mL]) | Baseline and up to 42 days
Part 3, Sub cohort 7: Number of participants with AEs, SAEs, and withdrawals due to AEs | Week 7 to 54 weeks
Part 3, Sub cohort 7: Number of participants with clinically significant changes in laboratory parameters and vital signs | Week 7 to 54 weeks
Part 4: Number of participants with HBsAg loss | Up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- Canada (2):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Ottawa, Ontario
- France (4):
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Rennes
- Italy (2):
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Monza MB
- South Korea (3):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
- GSK Investigational Site, Bangkok, Thailand
- United Kingdom (2):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com